CLINICAL TRIAL: NCT03544593
Title: The Volumetric Analysis of Fat Grafting for Aesthetic Body Contouring
Brief Title: The Volumetric Analysis of Fat Grafting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hunstad Kortesis Bharti Cosmetic Sugrery (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Bill G Kortesis, MD, PI, Hunstad Kortesis Bharti Cosmetic Sugrery
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 11-01-2017
Record Dates: First submitted 2018-05-08; First posted 2018-06-04 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Autologous Fat Grafting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Revolve System — Fat grafting system

SUMMARY:
Title: The Volumetric Analysis of Fat Grafting for Aesthetic Body Contouring.

Subjects who wish to undergo fat grafting for aesthetic body contouring will be offered enrollment to the study. The study will consist of a Screening/Baseline visit, Surgery day and 3 follow up visits. Each follow up visit will utilize Vectra 3D photography (Canfeild, NJ) to collect volumetric data. At the conclusion of the study, Volume data from Baseline and 3 follow up visits will be analyzed to determine fat retention rates.

ELIGIBILITY:
Inclusion Criteria:

1. Females or Males in good general health age 18 - 65 years of age
2. Must be willing to give and sign a HIPAA form and informed consent form
3. Must be willing and able to comply with all study protocols and schedules
4. Negative urine pregnancy test prior to surgery treatment (if applicable)
5. The patient must have had a stable weight (no fluctuation of >15 pounds in a year), diet, and physical activity for the previous 6 months

Exclusion Criteria:

1. Pregnancy, currently breast feeding or planning pregnancy for the duration of the trial
2. History of breast cancer if fat grafting to breasts
3. Patients who smoke or use nicotine products
4. Any UNCONTROLLED systemic disease -a potential patient in whom therapy for a systemic disease is not yet stabilized will not be considered for entry into the study
5. Diabetes Mellitus
6. Subject has a clinically significant coagulation disorder or disease, defined as a platelet count < 100,000 per microliter or International Normalized Ratio > 1.5 within 4 weeks of surgery
7. Patients under the age of 18
8. Patients undergoing fat grafting but refuse enrollment
9. Patients with an active infection
10. Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-01-04 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Graft retention | 9 months
  Vectra 3D volumetric analysis will be utilized to evaluate graft retention.

SECONDARY OUTCOMES:
Volume of adipose harvested (mL) | Intra Op
Volume of adipocyte injected (mL) | Intra Op
Operating room time (harvesting, processing, and reinjection time) (min) | Intra Op
Standardized before and after photos | Pre op, 3 months, 6 months, 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Costin, RN, BSN, Study Director — Hunstad Kortesis Bharti Cosmetic Surgery
Locations (1):
- Kelly Costin, Huntersville, North Carolina, United States